CLINICAL TRIAL: NCT03499418
Title: Evaluation of the Prevalence of Persistent Pulmonary Hypertension in Term and Near-term Neonates - Observational Study
Brief Title: Evaluation of the Prevalence of Persistent Pulmonary Hypertension in Neonates
Acronym: PRE-HIFREQ
Status: Withdrawn | Type: Observational
Why Stopped: Due to changing methodology of the study
Sponsor: Princess Anna Mazowiecka Hospital, Warsaw, Poland (Other)
Responsible Party: Principal Investigator, Renata Bokiniec, MD, Clinical Professor, Head of Department of Neonatology, Princess Anna Mazowiecka Hospital, Warsaw, Poland
Other Study IDs: PRE-HIFREQ
Record Dates: First submitted 2017-10-19; First posted 2018-04-17 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Transient Tachypnea of the Newborn; PPHN
Keywords: newborn; TTN; PPHN
MeSH Terms: conditions — Transient Tachypnea of the Newborn | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples Without DNA — blood gases
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- newborns with TTN: Group of late preterm and full-term newborns with TTN evaluated by modified Silverman scale
  Interventions: Other: modified Silverman scale
- newborns with PPHN: Group of late preterm and full-term newborns with respiratory failure with PPHN evaluated by echocardiography
  Interventions: Other: modified Silverman scale; Diagnostic Test: echocardiography

INTERVENTIONS:
Other: modified Silverman scale — Clinical assessment of severity of respiratory failure
Diagnostic Test: echocardiography — echocardiographic evaluation of haemodynamic problems
  Groups: newborns with PPHN

SUMMARY:
Transient Tachypnea of the Newborn (TTN) is one of the common causes of neonatal respiratory distress as a result of delayed clearance of fetal lung fluid.

Neonates with TTN usually require noninvasive respiratory support (e.g. nasal cannula, nasal CPAP) and may need supplemental oxygen therapy to maintain normal oxygen saturation levels. There have also been reports of "malignant TTN," in which affected children develop persistent pulmonary hypertension of the newborn (PPHN).

DETAILED DESCRIPTION:
Respiratory failure after birth is still a severe problem. Risk factors include premature labor and delivery by cesarean section. Despite the improvement of the quality of perinatal care in Poland, almost a constant percentage of premature babies has been born in Poland. The number of births by cesarean section is also rising - both planned and preceded by the attempt to vaginal delivery. TTN - Transient Tachypnea of the Newborn is one of the most common causes of respiratory failure in newborns. TTN occurs in approximately 10% of newborns born between 33 and 34 weeks of gestation, in about 5% of newborns born between 35 and 36 weeks and less than 1% of neonates.

At baseline of transient tachypnea of the newborn (TTN), there are disorders of absorption of pulmonary fluid. In the flow of water, epithelial sodium channels and Na+ / K+ -ATPase play an essential role. Their stimulation increases the absorption of water from the lung airspace and increases its transport both inside and outside the cell. In the subsequent stages of removal of interstitial pulmonary fluid, the vascular system and the lymphatic system are involved.

TTN is usually a self-limiting process, and treatments are not defined. There are also reports of "malignant TTN" in which infants develop persistent pulmonary hypertension of newborns (PPHN) (3). TTN infants typically require non-invasive respiratory support (CPAP, for example) and may need higher oxygen concentrations in the respiratory mixture to maintain proper oxygenation. Some experts suggest that the early use of expanding pressure (nasal CPAP) may relieve severe forms of TTN and prevent using of mechanical ventilation, and also may eventually prevent the development of persistent pulmonary hypertension.

Persistent pulmonary hypertension of newborns (PPHN) is a disorder arising at the stage of a physiological passage of fetal circulation into the neonatal circulation in the perinatal period. It is associated with a lack of decreasing pulmonary vascular resistance, which is influenced by increasing levels of oxygen in the blood and numerous biochemical and hormonal factors. From own observations and data from the literature, it is estimated that PPHN occurs in approximately 0.1-0.2% of newborns born term or near the term. Treatment of persistent pulmonary hypertension is difficult. Despite the use of mechanical ventilation, inhaled nitric oxide (iNO) or extracorporeal oxygenation (ECMO), the risk of death is still around 10-15%. This percentage has declined in recent years, but it is believed that persistent pulmonary hypertension of newborns is one of the most challenging situations in intensive care of newborns. In addition, infants who have undergone PPHN are exposed to long-term effects in the form of neurological complications or neurodevelopmental disorders.

Before initiating a clinical trial (intervention) with the experimental therapy, an initial follow-up study was conducted to assess the incidence of failure in respiratory insufficiency and the rate of PPHN in neonates born between 32 and 41 weeks of gestation. The failure of treatment will be defined as the need for invasive ventilation (intubation and mechanical ventilation). To accurately determine the degree of respiratory failure, a scale was developed that was an adaptation of the Silverman scale. PPHN will be defined by parameters measured in echocardiography and on changes in blood gases. Also, a comparison of parameters of acid-base balance and the type of treatment of respiratory failure after birth will be performed in the follow-up study. Based on the collected data, validation of the modified Silverman scale and evaluation of its clinical utility will be presented.

ELIGIBILITY:
Inclusion Criteria:

* A signed form of informed consent from parents (legal guardians).
* 32 0/7 to 41 6/7 weeks of gestation
* The need to support postnatal breathing, no later than 6 hours of life.

Exclusion Criteria:

* The need for intubation in the after-birth procedures
* Age above 6 hours of age from birth
* Congenital heart defects
* Congenital diaphragmatic hernia
* Other severe congenital malformations and genetically determined syndromes, diagnosed before and after birth, associated with higher risk of respiratory failure.

Ages: 10 Minutes to 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study is a multicenter, prospective, cohort, observational to assess the clinical benefits of using a scale in a population of neonates from 32 to 41 completed weeks PMA who will be admitted to a neonatal intensive care unit (NICU). Before study enrollment, parents (legal guardians) will provide a signed written informed consent form (ICF). ICF form may be signed after subject met inclusion criteria for the study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2023-03-31 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Rate of PPHN | 12 months
  The primary endpoint for this study is time of respiratory failure (need to intubation) and incidence rate of PPHN

SECONDARY OUTCOMES:
The evaluation of the "TTN scale" | 12 months
  The evaluation of the "TTN scale" in comparison to physiologic parameters:
  * Fraction of inspired oxygen (FiO2)
  * pH
  * Partial pressure of carbon dioxide (pCO2)

CONTACTS AND LOCATIONS:
Overall Officials: Maria K. Borszewska-Kornacka, MD, ProfTit, Study Chair — Medical University of Warsaw
Locations (1):
- Department of Neonatology and Neonatal Intensive Care Medical University of Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Raju TN, Higgins RD, Stark AR, Leveno KJ. Optimizing care and outcome for late-preterm (near-term) infants: a summary of the workshop sponsored by the National Institute of Child Health and Human Development. Pediatrics. 2006 Sep;118(3):1207-14. doi: 10.1542/peds.2006-0018. PMID 16951017
- [Background] Rubaltelli FF, Dani C, Reali MF, Bertini G, Wiechmann L, Tangucci M, Spagnolo A. Acute neonatal respiratory distress in Italy: a one-year prospective study. Italian Group of Neonatal Pneumology. Acta Paediatr. 1998 Dec;87(12):1261-8. doi: 10.1080/080352598750030951. PMID 9894827
- [Background] Lakshminrusimha S, Keszler M. Persistent Pulmonary Hypertension of the Newborn. Neoreviews. 2015 Dec;16(12):e680-e692. doi: 10.1542/neo.16-12-e680. PMID 26783388
- [Background] Buchiboyina A, Jasani B, Deshmukh M, Patole S. Strategies for managing transient tachypnoea of the newborn - a systematic review. J Matern Fetal Neonatal Med. 2017 Jul;30(13):1524-1532. doi: 10.1080/14767058.2016.1193143. Epub 2016 Oct 20. PMID 27762156